CLINICAL TRIAL: NCT02595606
Title: 0.3% Sodium Hyaluronate in the Treatment of Dry Eye of Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wang Zhichong, cornea department chief, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03SHDD
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Dry Eye Syndromes; Diabetes Mellitus
Keywords: dry eye syndromes; diabetes mellitus
MeSH Terms: conditions — Dry Eye Syndromes; Diabetes Mellitus | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment group (Experimental): treatment with 0.3% Sodium Hyaluronate, by five times a day, one or two drop each time
  Interventions: Drug: 0.3% Sodium Hyaluronate
- control group (No Intervention): without treatment

INTERVENTIONS:
Drug: 0.3% Sodium Hyaluronate — five times per day for the intervention of eye drop
  Arms: treatment group

SUMMARY:
A randomized parallel controlled study was designed to compare the efficacy of 0.3% Sodium Hyaluronate in the treatment of Dry Eye of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. medical history of diabetes
2. diagnosed with proliferative diabetic retinopathy
3. diagnosed with dry eye
4. not involvement in other drug experiment in the past 2 weeks
5. vision acuity better than 0.1
6. no local drug using history or with at least 2 weeks blanking period

Exclusion Criteria:

1. allergy to any of the drug ingredient
2. being or going to be pregnant or in lactation period
3. with any other eye disease or other serious disease which might affect the trial or could not get in follow-up
4. with any eye surgery history in the past six months
5. usage of hormone for replacement therapy

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
ocular surface disease index | up to 2 months
  pre-,1,4,8 weeks after the initiation of the study(the use of drug for experimental group)

SECONDARY OUTCOMES:
tear break up time | up to 2 months
  BUT
Schirmer' test | up to 2 months
  test of tear secretion
conjunctival goblet cells density | up to 2 months
  indirect assessment of tear quality
corneal fluorescein staining assessment | up to 2 months
  assessment of the corneal invasion

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Dogru M. Tear secretion and tear film function in insulin dependent diabetics. Br J Ophthalmol. 2000 Oct;84(10):1210. doi: 10.1136/bjo.84.10.1210. No abstract available. PMID 11004112
- [Background] Fujishima H, Shimazaki J, Yagi Y, Tsubota K. Improvement of corneal sensation and tear dynamics in diabetic patients by oral aldose reductase inhibitor, ONO-2235: a preliminary study. Cornea. 1996 Jul;15(4):368-75. doi: 10.1097/00003226-199607000-00006. PMID 8776562
- [Background] Zhivov A, Stachs O. Re: "Increased Langerhan cell density and corneal nerve damage in diabetic patients: Role of immune mechanisms in human diabetic neuropathy" by Tavakoli et al. Cont Lens Anterior Eye. 2011 Apr;34(2):98; author reply 99. doi: 10.1016/j.clae.2010.12.003. Epub 2011 Jan 6. No abstract available. PMID 21215678
- [Background] Maruyama K, Asai J, Ii M, Thorne T, Losordo DW, D'Amore PA. Decreased macrophage number and activation lead to reduced lymphatic vessel formation and contribute to impaired diabetic wound healing. Am J Pathol. 2007 Apr;170(4):1178-91. doi: 10.2353/ajpath.2007.060018. PMID 17392158
- [Background] Gao N, Yin J, Yoon GS, Mi QS, Yu FS. Dendritic cell-epithelium interplay is a determinant factor for corneal epithelial wound repair. Am J Pathol. 2011 Nov;179(5):2243-53. doi: 10.1016/j.ajpath.2011.07.050. Epub 2011 Sep 13. PMID 21924232
- [Background] Lu W, Ebihara N, Miyazaki K, Murakami A. Reduced expression of laminin-5 in corneal epithelial cells under high glucose condition. Cornea. 2006 Jan;25(1):61-7. doi: 10.1097/01.ico.0000179932.21104.3c. PMID 16331044